CLINICAL TRIAL: NCT00287352
Title: Double Blind Placebo Controlled Investigation of Amantadine for Retarding Weight Gain in First Episode Adlt Psychotic Subjects Beginning Therapy With Olanzapine.
Brief Title: Study of Amantadine for Weight Stabilization During Olanzapine Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Karen A. Graham, Msc, MD/Principal Investigator, University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F1D-MC-X273; GCRC 2235
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Psychotic Disorder; Schizophreniform Disorder; Schizophrenia; Schizoaffective Disorder; Mood Disorders With Psychotic Features
Keywords: First episode psychosis
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Olanzapine; Amantadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-Blind Treatment (Placebo Comparator): Olanzapine continuing with placebo
  Interventions: Drug: Olanzapine and placebo
- Olanzapine, Amantadine (Active Comparator): Standard combine with Amantadine
  Interventions: Drug: Olanzapine, Amantadine

INTERVENTIONS:
Drug: Olanzapine, Amantadine — Olanzapine continuing as clinically indicated, Amantadine 100 mg tid
  Arms: Olanzapine, Amantadine
Drug: Olanzapine and placebo — Olanzapine continuing as clinically indicated
  Arms: Double-Blind Treatment

SUMMARY:
Weight gain associated with antipsychotic medication use is a major side effect that limits the tolerability of these drugs. This often significant weight gain adversely affects health, increasing risks for developing cardiovascular disease, diabetes, sleep apnea, cancers of the colon, kidneys, uterus, endometrium and esophagus and osteoarthritis. Beasley and colleagues (1997) reported that 40.5% of olanzapine-treated patients gained more than 7% of baseline weight. Much of the olanzapine induced weight gain occurs early in treatment, and antipsychotic-naïve and young patients (Woods et al., 2002) are particularly vulnerable to this side effect. One of the most promising medications to aid weight loss in patients taking olanzapine is amantadine.

Attempts at preventing weight gain are expected to be more successful than attempts to reverse it once it occurs. It is now common clinical practice to educate all patients beginning treatment with olanzapine, and other antipsychotics, about healthy eating and the need for exercise. However, despite this effort, weight gain in this population continues. Beginning a weight-stabilizing medication after a low threshold of weight gain has occurred may have significant impact on patients' health and their willingness to continue to take antipsychotics.

We propose to investigate the efficacy of amantadine as a weight-stabilizing agent in a population of first-episode psychotic subjects just beginning treatment with antipsychotic agents. This population is generally young and medically healthy, without contraindications to amantadine. They are often of normal body mass index and without obesity-related medical problems. They have much to gain in preventing the weight gain which so often progresses steadily over the course of treatment, is difficult to reverse and results in significant morbidity and mortality. Additionally, the first episode psychotic population tends to take fewer concomitant psychiatric medications. This is important since these medications may cause weight gain (long term use of mirtazapine, lithium, depakote) or weight loss (short term use of SSRI's) which could confound the effectiveness of amantadine to combat weight gain.

DETAILED DESCRIPTION:
Screening: Screening will include demographics, medical and psychiatric histories and a clinical interview to determine psychiatric diagnosis. Screening will also include a physical examination and laboratory assessments (CBC, electrolytes, kidney function, liver function, TSH) to rule out concurrent medical illness that could be a contraindication to amantadine treatment. Blood will also be drawn for fasting lipid profile, glucose, insulin, C reactive protein, adiponectin, and leptin. Subjects will also have the option of allowing us to draw 2 additional tubes for as yet to be determined studies, not to include HIV or genetic testing. Subjects will also have the option of allowing us to draw 1 additional tube for platelet-specific protein assay, termed SEPT5. The rationale for measuring SEPT5 levels is to test a hypothesis that individuals with clinically-defined mental disorders have altered levels of this protein in their circulating blood platelets. A urine drug screen will be performed.

Phase 1: Subjects may enter Phase 1 within the first 12 weeks of treatment with olanzapine. At entry into Phase 1, anthropometric measurements will be taken (height, weight, waist and hip circumference) and BMI calculated. Baseline assessments will include questionnaires about hunger (to be done in the fasting state) (Subjective Satiety Scale), and activity (Baeckea Activity Questionnaire), respiratory quotient (RQ) and resting energy expenditure (REE) assessed using the Medgraphics metabolic cart, and body composition determined by dual x-ray absorptiometry (DXA, Hologic Delphia). Prior to every DXA scan Body Composition Lab personnel will administer a safety questionnaire and women of reproductive age will have a blood pregnancy test. Visits will be scheduled weekly to monitor weight and to provide healthy lifestyle counseling based on the Solutions for Wellness program developed by Lilly. During the first 3 weeks, subjects will be called by research personnel once per week to complete a 24 hour diet recall by phone. During the first 4 weeks of the study, RQ and capillary glucose will be repeated weekly since it is anticipated that changes to these parameters may occur early on. At monthly intervals clinical interviews will monitor for changes in psychosis and blood pressure will be assessed. When subjects gain 1 BMI unit, fasting bloodwork and baseline assessments are repeated and they are enrolled in Phase 2. Subjects who do not gain 1 BMI unit within 12 weeks of olanzapine treatment will end study participation at the end of Phase 1.

Phase 2: Subjects may enter Phase 2 following Phase 1 or enter directly if there is documentation of more than 1 but less than 3 BMI units of weight gain and they have started olanzapine within the previous 12 weeks. Phase 2 is a double blind placebo controlled addition of amantadine to ongoing olanzapine therapy. All subjects entering Phase 2 will have anthropometric measurements, and BMI will be calculated. Fasting lipid profile, glucose, insulin, C reactive protein, adiponectin, and leptin will be obtained, as will liver function tests and a urine drug screen. Body composition by DXA as well as RQ and REE will be determined. Prior to every DXA scan the Body Composition Lab will administer a safety questionnaire and women of reproductive age will have a pregnancy test. A Food Propensity questionnaire will be administered to document recent trends in food choices, and the exercise and hunger questionnaires will also been done. Following completion of baseline assessments, randomization to amantadine or placebo will occur. Subjects will begin taking 1 capsule daily for 2 days, 2 capsules daily for 5 days, and then 3 capsules daily. Amantadine capsules will each contain 100 mg of amantadine. Clinical state and emergence of side effects, including orthostatic hypotension, will be monitored at all visits by research clinicians. If subjects experience mild side effects with increase in number of capsules, the titration will be slowed. During Phase 2, subjects will be called by research personnel on 3 nonconsecutive days to complete a 24 hour diet recall by phone. Biweekly, all subjects will meet with a study physician or nurse for standardized healthy lifestyle counseling based on the Solutions for Wellness program available from Lilly. BMI will be calculated biweekly and baseline measures will be repeated at the final study visit. Urine pregnancy test will be performed monthly on all women. When subjects gain an additional 3 BMI units (approximately 15 lbs), or when they complete 16 weeks of double blind medication they will repeat all Visit 13 measures and end study participation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Male and female
* DSM IV diagnosis of psychotic episode (brief psychotic disorder, schizophreniform disorder, schizophrenia, schizoaffective disorder)or mood disorder with psychotic features
* Subjects may have lifetime exposure to antipsychotic medications other than olanzapine of up to 8 weeks
* Olanzapine monotherapy is appropriate treatment as judged by their treating physician.

Less than 12 weeks of olanzapine monotherapy treatment at entrance into phase 1.

* Able to consent
* Female subjects require medically acceptable means of birth control which includes tubal ligation, hysterectomy, condoms, oral contraceptives, IUD, cervical cap, diaphragm, transdermal contraceptive patch, and abstinence.

Exclusion Criteria:

* Current treatment with lithium, depakote, carbamazepine, lamotrigine, mirtazapine, corticosteroids, or stimulants (methamphetamine, etc).
* Known sensitivity or contraindication to amantadine
* Suicidal or homicidal risk
* Pregnant, desiring to become pregnant during the study period, or lactating
* Serious or unstable medical illness that require ongoing treatment with medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare time to clinical significant weight gain in the amantadine + olanzapine group with the placebo + olanzapine group. | 29 weeks

SECONDARY OUTCOMES:
We will determine if the amantadine + olanzapine group has a lower % body fat compared to the placebo + olanzapine group at 16 weeks | 29 weeks
We will determine if the amantadine +olanzapine group has a higher RQ signifying better fat utilization compared to the placebo + olanzapine group at 16 weeks | 29 weeks
We will determine if the amantadine + olanzapine group has significantly better metabolic profile at 16 weeks as compared to the placebo + olanzapine group. | 29 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Graham, MSc MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States